CLINICAL TRIAL: NCT04700605
Title: Intra-rater Reliability and Agreement Between Static Balance Test Using Nintendo Wii Balance Board and Gait Test Under Dual Task Conditions in Community-dwelling Older Adults.
Brief Title: Intra-rater Reliability and Agreement Between Two Dual Task Tests; WBB and Gait Test.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Martin Eriksen, Medical student, Aalborg University Hospital
Other Study IDs: 2020-096
Record Dates: First submitted 2021-01-04; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Balance; Distorted

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Dual task balance test — Participants will be conducting two dual task tests; an 8m gait test and a Wii Balance Board test with simultaneous various cognitive tests.

SUMMARY:
Agreement and intra-rater reliability between static balance test using Nintendo Wii Balance Board and gait test under dual-task conditions in community-dwelling older adults.

DETAILED DESCRIPTION:
Participants:

Investigators aim to recruit a minimum of 30 participants aged 65 years or above through convenience sampling at an senior activity centre in the Municipality of Aalborg. Participants inclusion critiria is age about 65, the ability to stand for 30 seconds unaided and the ability to walk 8 meters. Exclusion critiria is severe cognitive impairment (e.g., dementia).

Procedure:

Each participant will undergo two testdays separated by approximately two weeks. Both testdays have the same number and order of tests and are placed approximately the same time of the day. At the first testday descriptive information for each participant is collected.

Measuring device:

The Nintendo Wii Balance Board (Nintendo, Kyoto, Japan) is a small portable force plate measuring sway ellipse area and sway speed.

Analysis:

Will include intra-rater reliability for each test and agreement between the two. Calculations of balance/gait costs will be made to unify the unit and to compare the two tests to each other. Results shown by intraclass correlation coeffients and Bland Altman plots.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 65 years old.
* Community dwelling

Exclusion Criteria:

* Unable to stand unsupported for 30 seconds
* Unable to walk 8 meters unsupported

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Minimum 65 year-old community dwelling citizens at activity centers.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-01-06 (Estimated); Study Completion 2021-01-06 (Estimated)

PRIMARY OUTCOMES:
Intra-rater reliability for the gait test and the WBB test. | Through study completion, app. 8 months.
  Comparing the dual task costs for each test between test and retest. Assessments through intraclass correlation coefficient and reportings in accordance with Guidelines for Reporting Reliability and Agreement Studies (GRRAS).

SECONDARY OUTCOMES:
Agreement between the gait test and the WBB test as dual task measurements. | Through study completion, app. 8 months.
  Comparing the dual task costs between the gait test and the Wii Balance Board test. Data assessment through Bland Altman plots and reportings in accordance with Guidelines for Reporting Reliability and Agreement Studies (GRRAS).
Descriptive data. | Through study completion, app. 8 months.
  Qustionnairies consisting of Tilburg Frailty Indicator, Vulnerable Elders Survey 13, Short Falls Efficacy Scale, previous falls, medications and Orientations-Memory-Concentrations test. Data assessment through histograms and Shapiro Wilk tests and reported by means and standard deviations, medians and interquartile ranges, and numbers and percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Eriksen, Principal Investigator — Aalborg University Hospital
Locations (1):
- Liselund Aktivitets Center, Vodskov, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT04700605/Prot_000.pdf